CLINICAL TRIAL: NCT05353322
Title: Breaking up Prolonged Sedentary Behavior to Improve Cardiometabolic Health: An Adaptive Dose-Finding Study
Brief Title: Breaking up Prolonged Sedentary Behavior to Improve Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Keith Diaz, Associate Professor of Behavioral Medicine, Columbia University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: AAAT9416; 1R01HL153642-01A1 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Sedentary Behavior; Cardiometabolic Risk Factors; Blood Pressure; Glucose
Keywords: Sedentary Behavior; Physical Activity; Blood Pressure; Glucose; Insulin; Dose-finding
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Insulin Resistance | interventions — Walking; Sitting Position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedentary Break Condition > Control Condition (Experimental): Participants will be assigned to the sedentary break or control condition at each lab visit. If assigned to the sedentary break condition at lab visit 1, participants will be assigned to the control condition at visit 2 (and vice versa). During the lab visit, participants will wear a heart rate monitor and ambulatory blood pressure monitor, and eat a controlled diet. Participants will also eat a controlled diet for two days prior to the lab visit.
  Interventions: Behavioral: Sedentary Break (Walking) Condition; Behavioral: Sitting (Control) Condition; Behavioral: Controlled Diet
- Control Condition > Sedentary Break Condition (Experimental): Participants will be assigned to the sedentary break or control condition at each lab visit. If assigned to the sedentary break condition at lab visit 1, participants will be assigned to the control condition at visit 2 (and vice versa). During the lab visit, participants will wear a heart rate monitor and ambulatory blood pressure monitor, and eat a controlled diet. Participants will also eat a controlled diet for two days prior to the lab visit.
  Interventions: Behavioral: Sedentary Break (Walking) Condition; Behavioral: Sitting (Control) Condition; Behavioral: Controlled Diet

INTERVENTIONS:
Behavioral: Sedentary Break (Walking) Condition — For the sedentary break (walking) condition, participants will be randomized to 1 of 25 combinations of frequency (5 doses: sedentary break every 30, 45, 60, 90, or 120 minutes) and duration (5 doses: sedentary break duration of 1, 3, 5, 7, or 10 minutes). Participants will complete a 9-hour study visit and will remain seated throughout the lab visit and will take regular sedentary breaks by walking on a treadmill at 2.0 mph and 0% incline at specific frequency and duration (as determined by the randomization method) for the entirety of the visit.
  Other Names: Sedentary Break (Walking) Condition - Experimental
Behavioral: Sitting (Control) Condition — While completing the sitting (control) condition, participants will complete the 9-hour study visit by remaining seated and only standing up/walking to use the restroom at specified times.
  Other Names: Sitting (Control) Condition - Shame Comparator
Behavioral: Controlled Diet — Participants in both the experimental and control groups will eat a controlled diet (breakfast, lunch, dinner, snacks) for two full days before each lab visit. They will also eat a controlled diet (breakfast, lunch) during each of the two lab visits. Participants will choose 1 of 3 dietary menus to eat for the study duration. Each meal will be individualized to meet 33% of daily estimated energy requirements. Target macronutrient profile will be 12-15% energy from protein, 55-58% from carbohydrate and 29-31% from fat; as well as 55 mmol of sodium and 24 mmol of potassium.
  Other Names: Controlled Foods Diet

SUMMARY:
The purpose of this Phase 1 research study is to answer two questions: (1) How frequent should periods of prolonged sedentary time be interrupted? and (2) What is the appropriate duration or length of time of these breaks in sedentary time? To address these questions, this project will conduct a state-of-the-art adaptive dose finding study under controlled laboratory conditions to determine the minimally effective dose (the smallest dose) that yields cardiometabolic benefit for two separate sedentary break elements (frequency and duration). Study findings will ultimately determine how often and for how long people should break up periods of prolonged sedentary time to transiently improve established cardiovascular risk factors; key foundational information critical to the success of future long-term trials and ultimately public health guidelines.

Primary Aim: To determine the minimally effective dose combination(s) of frequency and duration needed to provide cardiometabolic benefit during an 8-hour experimentation period. Specifically, the study will determine:

1a. For each fixed duration, the minimum sedentary break frequency (e.g., every 30 min, 60 min, 120 min) that demonstrates a reduction in systolic BP, diastolic BP, or glucose compared with a sedentary control condition.

1b. For each fixed frequency, the minimum sedentary break duration (e.g., activity breaks of 1 min, 5 min, 10 min) that demonstrates a reduction in systolic BP, diastolic BP, or glucose compared with a sedentary control.

Secondary Aim: It is also critical to public health strategy to assess the acceptability/feasibility of various sedentary break doses as too high a dose will yield poor uptake. To address this need, the maximally tolerated dose (the highest dose that does not cause undue physical/psychological distress) for frequency and duration of sedentary breaks will also be determined via assessment of 4 constructs: physical exhaustion/fatigue, affect (e.g., mood, emotion), tolerability (e.g., completion of dose protocol), and safety (e.g., hypoglycemia). Maximally tolerated dose will be defined as the highest dose where <20% of participants exhibit an adverse outcome.

DETAILED DESCRIPTION:
Excessive sedentary behavior is highly prevalent in developed nations and is a risk factor for cardiovascular disease (CVD) morbidity and mortality. Evidence suggests sedentary behavior is not simply a form of inactivity that elicits positive energy balance. Instead sedentary behavior itself may be harmful. As such, health agencies have provided general recommendations to "sit less, move more" by interspersing brief periods of activity. However, a lack of empirical evidence describing how often (e.g. every 30 min, every 60 min) and for how long (e.g. 1 min activity bouts, 5 min activity bouts) sedentary time should be interrupted (a "sedentary break") to yield health benefit has precluded more quantitative, actionable guidelines. To date, rigorous and methodical dose escalation experiments have not been conducted to elucidate efficacious and tolerated sedentary break doses. Without specific targets to provide to the public; public health initiatives targeting sedentary behavior will likely have minimal effectiveness. Critically, without rigorously tested dosing information; randomized controlled trials targeting sedentary behavior may be fruitless; bearing risk of inefficacious or intolerable doses. The objective of the proposed study is to determine the minimally effective dose (e.g. the smallest dose) for two elements of a sedentary break, frequency and duration, that yields improvements in established CVD risk factors. The investigator will also determine the maximally tolerated dose (e.g. the highest dose that does not cause undue physical/psychological distress) for both frequency and duration of sedentary breaks. To address the aims, the investigator will conduct a state-of-the-art dose finding study under well controlled laboratory conditions using an innovative Bayesian adaptive randomization method for dose determination never before applied to behavioral trials. This method will enable us to efficiently test 25 possible frequency/duration combinations in just a single study. The study will recruit 324 adults to complete a total of 2 trial conditions in the laboratory (8 hours each), namely a sedentary break (active) condition and an uninterrupted sitting (control) condition, in a randomized order. The sedentary break condition will consist of 1 of 25 possible frequency/duration combinations (e.g. every 30 min for 10 min), selected according to the adaptive randomization protocol. Established CVD risk factors, including blood pressure and glucose, as well as measures of dose tolerability (physical exhaustion/fatigue, affect) and work engagement and performance will be serially assessed during each trial.

This project is a groundbreaking step towards developing evidence-based guidelines for sedentary behavior that will establish a foundation upon which a successful sedentary behavior intervention development process can be rooted. By identifying the minimally effective and maximally tolerated dose combinations for the frequency and duration of a sedentary break; this Phase I/II study will provide key foundational evidence critical to the success of future Phase III and Phase IV randomized trials and ultimately public health guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to read, write and speak English or Spanish
* Limited or no chronic medical conditions [examples include but not limited to: CVD, diabetes, chronic obstructive pulmonary disease (COPD), HIV/AIDS; participants with high blood pressure/hypertension and/or high cholesterol/hyperlipidemia may be included if they are currently prescribed and taking medication for these conditions]
* Do not take medication (over-the-counter or herbal) to control glucose (such as a diabetes control medication)
* Not currently pregnant
* Do not currently smoke cigarettes
* No pre-existing musculoskeletal conditions (including but not limited to osteoarthritis, rheumatoid arthritis, psoriatic arthritis, gout, ankylosing spondylitis) that would prevent participation in intermittent physical activity
* No allergies to common food allergens including wheat, eggs, milk or other dairy, gluten, fructose, peanuts or other nuts
* No dietary restrictions such as vegan, gluten free, halal

Exclusion Criteria:

• Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure from Baseline | Baseline, 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 5.5 hours, 6 hours, 6.5 hours, 7 hours, 7.5 hours, 8 hours
  Measured by Spacelabs 90227 Ambulatory Blood Pressure Monitor and appropriately sized cuff on the non-dominant arm. Measured every 30 minutes over 8-hour trial visit (total of 18 individual readings).
Change in Diastolic Blood Pressure from Baseline | Baseline, 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 5.5 hours, 6 hours, 6.5 hours, 7 hours, 7.5 hours, 8 hours
  Measured by Spacelabs 90227 Ambulatory Blood Pressure Monitor and appropriately sized cuff on the non-dominant arm. Measured every 30 minutes over 8-hour trial visit (total of 18 individual readings).
Net Glucose Incremental Area Under the Curve | Every 15 minutes over 8-hour trial visit
  Interstitial glucose levels are measured every 15 minutes over 8-hour trial visit using the Freestyle Libre Pro Continuous Glucose Monitor inserted on deltoid of the dominant arm.

SECONDARY OUTCOMES:
Proportion of participants that fully completed the sedentary break protocol. | Immediately after completion of experimental (activity break) trial visit (up to 8 hours)
  This is to measure intervention tolerability. Tolerability is defined as full completion of the sedentary break protocol. That is, if the sedentary break dose is every 60 min for 5 min (a total of 40 min of activity over the 8 hour visit); the participant is able walk for a full 5 min every 60 min (thus walking 40 out of a possible 40 min).
Proportion of participants with hypoglycemia | Baseline, 0.5 hour, 1 hour, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours
  Hypoglycemia is defined as glucose levels <70 mg/dL. For each sedentary break dose, the study will calculate the proportion of participants who exhibit hypoglycemia based off serially measured blood glucose levels.
Proportion of participants with an exaggerated blood pressure response | Baseline, 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 4.5 hours, 5 hours, 5.5 hours, 6 hours, 6.5 hours, 7 hours, 7.5 hours, 8 hours
  An exaggerated blood pressure response is defined as systolic blood pressure ≥210 mm Hg for men and ≥190 mm Hg for women. For each sedentary break dose, the study will calculate the proportion of participants with an exaggerated blood pressure response based off of serially collected blood pressure measurements.
Proportion of participants in whom a musculoskeletal injury was observed/reported. | End of experimental (activity break) trial visit (up to 8 hours)
  This is to measure the prevalence of musculoskeletal Injury. Observed by research coordinator or self-reported by participant. For each sedentary break dose, the study will calculate the proportion from the collected data.
Proportion of participants reporting physical exhaustion score greater than or equal to 9 | Baseline, 4 hours, 8 hours
  This is to measure strong feelings of fatigue/exhaustion. The Physical Exhaustion Subscale of the Exercise-Induced Feeling Inventory consists of 3 exhaustion/fatigued-related items ("Fatigued", "Tired", "Worn-out") and response options on a 5-point scale from 0 (do not feel) to 4 (feel very strongly). Responses are summed with higher scores indicating greater perceived physical exhaustion.
Proportion of participants reporting Feeling Scale Score less than 0 | Up to 8 hours
  This is to measure negative affective valence. The Feeling Scale is single-item questionnaire which measures pleasure/displeasure in response to physical activity. Participants are asked to rate their present feelings on an 11-point good/bad bipolar scale from -5 (very bad) to +5 (very good).
Blood Insulin Area Under the Curve | Baseline, 0.5 hour, 1 hour, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours
  Blood samples are serially collected ten times over 8-hour trial visit by intravenous catheter. Insulin is assayed in duplicate.
Blood Glucose Area Under the Curve | Baseline, 0.5 hour, 1 hour, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours, 8 hours
  Blood samples are serially collected ten times over 8-hour trial visit by intravenous catheter. Glucose is assayed in duplicate.

OTHER OUTCOMES:
Utrecht Work Engagement Scale (UWES-9) Score | 4 hours, 8 hours
  Work Engagement - Measured by the Utrecht Work Engagement Scale (UWES-9) Score, adapted for momentary administration. The UWES-9 evaluates three dimensions of work engagement - vigor, dedication, and absorption - using a 7-point Likert scale. Higher scores reflect higher work engagement.
Work Performance Score | 4 hours, 8 hours
  Perceived work performance quantity and quality, along with an overall rating of work performance, will be measured by the World Health Organization Health and Work Performance Questionnaire (HPQ), adapted for momentary administration. The HPQ includes two items that measure performance quantity (e.g. ""How often did you not work at times when you were supposed to be working") and three items that measure performance quality on a 5-point Likert scale; along with an overall rating of work performance on a 0 to 10 scale. Higher scores reflect higher perceived work performance.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Diaz, PhD, Principal Investigator — Florence Irving Assistant Professor of Behavioral Medicine, CUIMC; Ying Kuen (Ken) Cheung, PhD, Study Chair — Professor of Biostatistics, Department of Biostatistics, CUIMC
Locations (1):
- Center for Behavioral Cardiovascular Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz KM, Murdock ME, Clark AW, Kumar S, Jerez V, Serafini MA, Xu C, Boudreaux BD, Romero EK, Aguirre J, Seid H, Nandakumar R, Ginsberg H, Shimbo D, Cheung YK. Breaking up prolonged sedentary behavior to improve cardiometabolic health (BREAK2): protocol for a dose-finding adaptive randomization trial. BMC Public Health. 2025 May 25;25(1):1929. doi: 10.1186/s12889-025-22250-0. PMID 40414835